CLINICAL TRIAL: NCT03647449
Title: Examining the Effects of Juice Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Melinda Ring, Clinical Associate Professor of Medicine and Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00206611
Record Dates: First submitted 2018-07-16; First posted 2018-08-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Epigenetics; Microbiome
Keywords: Juice fasting; methylation; microbiome; caloric restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Juice fast (Experimental): In the "juice fasting" arm, participants will be given vegetable/fruit pressed juices and be instructed to engage in a three-day juice fast diet totaling 800-900 kcal-per-day. The specific juices will be assigned for each day in order to maintain the calorie level.
  Interventions: Dietary Supplement: Juice; Behavioral: Caloric restriction via Plant-based meals
- Caloric restriction via Plant-based meals (Experimental): In the "caloric restriction diet" arm, participants will be on a whole-food plant-based diet totaling 800-900 kcal-per-day (matching the daily calories of juice fasting).
  Interventions: Behavioral: Caloric restriction via Plant-based meals; Dietary Supplement: Plant-based meal
- Juice plus ad hoc (Experimental): In the "juice plus ad hoc" arm, participants will be given the same juice for three days but continue with their usual diet in addition to the juice. For this arm, there is no restriction of caloric intake or restriction to liquid only.
  Interventions: Dietary Supplement: Juice

INTERVENTIONS:
Dietary Supplement: Juice — Participants will be drinking 800-900 kcal/day in cold-pressed juices.
  Arms: Juice fast; Juice plus ad hoc
Behavioral: Caloric restriction via Plant-based meals — Participants' caloric intake will be limited to 800-900 kcal/day.
  Arms: Caloric restriction via Plant-based meals; Juice fast
Dietary Supplement: Plant-based meal — Participants will be eating ~900 kcal/day in pre-prepared plant-based meals.
  Arms: Caloric restriction via Plant-based meals

SUMMARY:
This study tests the effectiveness of dietary interventions that have the possibility to improve markers of gut health and improve general well-being. This study will allow healthcare professionals to learn how dietary interventions involving fasting can affect health. Food is increasingly recognized as a core component of preventive and ameliorative health care. Juice fasting has quickly become one of the most popular self-prescribed dietary interventions in the United States. A wide variety of juice fasts are available in the popular market; a popular variation is the three-day juice fast. The purpose of this study is to assess the effects of a three-day juice fast on certain markers of age-related disease and bio-markers of longevity. In particular, this study will assess certain epigenetic markers, which measure how the environment (including diet) can change the way that genes are expressed without changing the genes themselves. The study will also assess the microbiome, and inflammatory and glycemic markers.

DETAILED DESCRIPTION:
Up to 30 participants will be enrolled in the study and will be randomized into one of the three arms: the "juice fasting" arm, the "juice plus ad hoc" arm, and the "caloric restriction" arm. Participants will come into the lab for an initial visit, during which they will complete questionnaires on their usual diet and demographics and will be informed about their assignment to one of the three arms.

In all three arms, the three-day diet intervention will be preceded and followed by three days of self-conducted elimination diet. The pre-intervention diet will encourage participants to eat a healthy, light diet for three days (basic instructions: eat only fresh raw or cooked fruits and vegetables (preferably organic), whole grains and eggs; drink 8 glasses of water a day; avoid or eliminate alcohol, caffeine, sugar, processed foods, dairy, red meat, and gluten). The post- intervention diet will instruct participants to gradually return to eating solid foods, and limit strenuous exercise (basic instructions: follow a diet similar to the pre-intervention elimination diet; day 1 after the intervention: eat fruits & green vegetables, and drink 8 glasses of water; day 2 add in: nuts, gluten-free grains like whole oats, quinoa, or brown rice; day 3 add in: organic meats, fish, & gluten-containing grains).

Biological samples and self-reported outcomes will be collected at four time points: baseline (prior to the first elimination diet period), pre-intervention (after the elimination diet and before the three-day intervention), post-intervention (after the intervention), and 14-day post- intervention. At each time point, participants will complete questionnaire on quality of life (PROMIS - Global Health Scale, which is an NIH measure on an individual's' overall physical and psychological well-being; see appendix) and collect their stool samples. Participants will be provided self-administered tool kits and be taught how to collect the stool sample at their first lab visit. At each of the four time points, the research assistant will coordinate the collection of cheek swabs, saliva samples, and blood spot samples. Biometrics will also be collected at each time point (weight, waist circumference, and blood pressure).

Over the course of the study, participants will be instructed to keep a diet diary days one through nine to record their daily dietary intake. During the intervention period, the research team will also contact the participants for daily check-ins. Participants will not need to record diet data for the remaining 11 days of the post-intervention period.

At the conclusion of the study, participants will bring back the final biological samples (stool wipe and saliva), provide the set of samples, and be debriefed about the purposes of the study.

The biological samples collected will then be processed and assayed for microbiome, methylation, inflammatory markers, and glycemic markers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects considered as healthy by the investigator based on medical history and completion of the screening questionnaire.
* Subjects who, according to the investigator, can and will comply with the requirements of the protocol and are available for all scheduled visits at the investigational site.
* Healthy male or female aged between 18 and 35 (included) years
* 18.5 ≤BMI ≤ 30 kg/m²
* Ability to give their informed consent in writing

Exclusion Criteria:

* Documented history of previous cardiovascular disease, including coronary heart disease (CHD) (angina, myocardial infarction, coronary revascularization procedures or existence of abnormal Q waves in the electrocardiogram (EKG)), stroke, syncope, and clinical peripheral artery disease with symptoms of intermittent claudication.
* Severe medical condition that may impair the ability of the person to participate in a nutrition intervention study (e.g. digestive disease with fat intolerance, advanced malignancy, or major neurological, psychiatric or endocrine disease including diabetes).
* Daily use of any prescription or non-prescription medication that has a high likelihood of impacting systemic inflammation (e.g. non-steroidal anti inflammatories or steroids), blood sugar control (e.g. medication for diabetes) or the human microbiome (e.g. antibiotics).
* Any other medical condition thought to limit survival to less than 1 year.
* Known immunodeficiency disorder
* Illegal drug use or chronic alcoholism or total daily alcohol intake >80 g/d.
* Difficulties or major inconvenience to change dietary habits
* Impossibility to follow an elimination or juice fast diet, for religious reasons or due to the presence of disorders of chewing or swallowing (e.g., difficulties to consume nuts)
* A low predicted likelihood to change dietary habits according to the Prochaska and DiClemente stages of change model (Nigg, 1999).
* History of food allergy with hypersensitivity to any of the components of the juice or diet
* Patients with an acute infection or inflammation (e.g., pneumonia) are allowed to participate in the study 3 months after the resolution of their condition.
* Dietary restrictions due to medical (including allergies), religious, or other concerns
* Any diagnosis of allergic rhinitis, eczema, asthma, or inflammatory bowel disease (e.g. ulcerative colitis or Crohn's) from a health professional

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change DNA Methylation at Day 7 | This outcome will be measured on day 7 of the study.
  The ratio of methylated signal to total signal and the M-value (log2 ratio of methylated signal over unmethylated signal) will be determined for each interrogated locus using Illumina's Infinium Methylation EPIC BeadChip

SECONDARY OUTCOMES:
Baseline DNA Methylation | This outcome will be measured on day 1 of the study.
  The ratio of methylated signal to total signal and the M-value (log2 ratio of methylated signal over unmethylated signal) will be determined for each interrogated locus using Illumina's Infinium Methylation EPIC BeadChip
Change DNA Methylation at Day 4 | This outcome will be measured on day 4 of the study.
  The ratio of methylated signal to total signal and the M-value (log2 ratio of methylated signal over unmethylated signal) will be determined for each interrogated locus using Illumina's Infinium Methylation EPIC BeadChip
Change DNA Methylation at Day 21 | This outcome will be measured on day 21 of the study.
  The ratio of methylated signal to total signal and the M-value (log2 ratio of methylated signal over unmethylated signal) will be determined for each interrogated locus using Illumina's Infinium Methylation EPIC BeadChip
PROMIS Global Health self-report | This outcome will be measured on day 1 of the study.
  The PROMIS Global Health measures assess an individual's physical, mental, and social health. The measures are generic, rather than disease-specific, and often use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. and psychological well-being
PROMIS Global Health self-report, repeatable | This outcome will be measured on day 4 of the study.
  The PROMIS Global Health self-report, described in Outcome 5, will be administered daily during the active portion of the study.
PROMIS Global Health self-report, repeatable | This outcome will be measured on day 5 of the study.
  The PROMIS Global Health self-report, described in Outcome 5, will be administered daily during the active portion of the study.
PROMIS Global Health self-report, repeatable | This outcome will be measured on day 6 of the study.
  The PROMIS Global Health self-report, described in Outcome 5, will be administered daily during the active portion of the study.
Baseline Blood Pressure | This outcome will be measured on day 1 of the study.
  The investigators will measure systolic and diastolic blood pressure, which will be measured manually using a stethoscope and blood pressure cuff.
Blood Pressure at Day 4 | This outcome will be measured on day 4 of the study.
  The investigators will measure systolic and diastolic blood pressure, which will be measured manually using a stethoscope and blood pressure cuff.
Change in Blood Pressure at Day 7 | This outcome will be measured on day 7 of the study.
  The investigators will measure systolic and diastolic blood pressure, which will be measured manually using a stethoscope and blood pressure cuff.
Change in Blood Pressure at Day 21 | This outcome will be measured on day 21 of the study.
  The investigators will measure systolic and diastolic blood pressure, which will be measured manually using a stethoscope and blood pressure cuff.
Baseline Waist Circumference | This outcome will be measured on day 1 of the study.
  Waist circumference will be measured according to CDC guidelines: the participant will stand, and a tape measure will be placed horizontally around their middle, just above the hip bones.
Waist Circumference at Day 4 | This outcome will be measured on day 4 of the study.
  Waist circumference will be measured according to CDC guidelines: the participant will stand, and a tape measure will be placed horizontally around their middle, just above the hip bones.
Change in Waist Circumference at Day 7 | This outcome will be measured on day 7 of the study.
  Waist circumference will be measured according to CDC guidelines: the participant will stand, and a tape measure will be placed horizontally around their middle, just above the hip bones.
Change in Waist Circumference at Day 21 | This outcome will be measured on day 21 of the study.
  Waist circumference will be measured according to CDC guidelines: the participant will stand, and a tape measure will be placed horizontally around their middle, just above the hip bones.
Baseline Weight | This outcome will be measured on day 1 of the study.
  Weight will be measured using a digital scale and recorded in pounds
Weight at Day 4 | This outcome will be measured on day 4 of the study.
  Weight will be measured using a digital scale and recorded in pounds
Change in Weight at Day 7 | This outcome will be measured on day 7 of the study.
  Weight will be measured using a digital scale and recorded in pounds
Change in Weight at Day 21 | This outcome will be measured on day 21 of the study.
  Weight will be measured using a digital scale and recorded in pounds
Baseline C-Reactive Protein | This outcome will be measured on day 1 of the study
  C-reactive protein (CRP) is a blood test marker for inflammation in the body.
C-Reactive Protein at Day 4 | This outcome will be measured on day 4 of the study
  C-reactive protein (CRP) is a blood test marker for inflammation in the body.
Change in C-Reactive Protein at Day 7 | This outcome will be measured on day 7 of the study
  C-reactive protein (CRP) is a blood test marker for inflammation in the body.
Change in C-Reactive Protein at Day 21 | This outcome will be measured on day 21 of the study
  C-reactive protein (CRP) is a blood test marker for inflammation in the body.
Baseline Interleukin-6 | This outcome will be measured on day 1 of the study.
  Interleukin-6 (IL-6) is an endogenous chemical which is active in inflammation, and in B cell maturation. Besides being an immune protein, it is also a pyrogen, and is responsible for fever in autoimmune, infectious or non-infectious disease.
Interleukin-6 at Day 4 | This outcome will be measured on day 4 of the study.
  Interleukin-6 (IL-6) is an endogenous chemical which is active in inflammation, and in B cell maturation. Besides being an immune protein, it is also a pyrogen, and is responsible for fever in autoimmune, infectious or non-infectious disease.
Change in Interleukin-6 at Day 7 | This outcome will be measured on day 7 of the study.
  Interleukin-6 (IL-6) is an endogenous chemical which is active in inflammation, and in B cell maturation. Besides being an immune protein, it is also a pyrogen, and is responsible for fever in autoimmune, infectious or non-infectious disease.
Change in Interleukin-6 at Day 21 | This outcome will be measured on day 21 of the study.
  Interleukin-6 (IL-6) is an endogenous chemical which is active in inflammation, and in B cell maturation. Besides being an immune protein, it is also a pyrogen, and is responsible for fever in autoimmune, infectious or non-infectious disease.
Baseline Insulin Level | This outcome will be measured on day 1 of the study.
  A fasting insulin test will show fasting blood sugar levels.
Insulin Level at Day 4 | This outcome will be measured on day 4 of the study.
  A fasting insulin test will show fasting blood sugar levels.
Change in Insulin Level at Day 7 | This outcome will be measured on day 7 of the study.
  A fasting insulin test will show fasting blood sugar levels.
Change in Insulin Level at Day 21 | This outcome will be measured on day 21 of the study.
  A fasting insulin test will show fasting blood sugar levels.
Baseline Leptin | This outcome will be measured on day 1 of the study.
  Leptin is an adipocyte-derived hormone that is essential for normal body weight regulation. Leptin production is under neuroendocrine control so that serum concentrations vary directly with the amount of triglycerides stored in adipose tissue depots.
Leptin at Day 4 | This outcome will be measured on day 4 of the study.
  Leptin is an adipocyte-derived hormone that is essential for normal body weight regulation. Leptin production is under neuroendocrine control so that serum concentrations vary directly with the amount of triglycerides stored in adipose tissue depots.
Change in Leptin at Day 7 | This outcome will be measured on day 7 of the study.
  Leptin is an adipocyte-derived hormone that is essential for normal body weight regulation. Leptin production is under neuroendocrine control so that serum concentrations vary directly with the amount of triglycerides stored in adipose tissue depots.
Change in Leptin at Day 21 | This outcome will be measured on day 21 of the study.
  Leptin is an adipocyte-derived hormone that is essential for normal body weight regulation. Leptin production is under neuroendocrine control so that serum concentrations vary directly with the amount of triglycerides stored in adipose tissue depots.
Baseline Gut microbiota | This outcome will be measured on day 1 of the study.
  16S rRNA amplicon library created for taxonomic annotation analysis.
Gut microbiota at Day 4 | This outcome will be measured on day 4 of the study.
  16S rRNA amplicon library created for taxonomic annotation analysis.
Change in Gut microbiota at Day 7 | This outcome will be measured on day 7 of the study.
  16S rRNA amplicon library created for taxonomic annotation analysis.
Change in Gut microbiota at Day 21 | This outcome will be measured on day 21 of the study.
  16S rRNA amplicon library created for taxonomic annotation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Ring, MD, FACP, Principal Investigator — Osher Center for Integrative Medicine at Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Redman LM, Ravussin E. Caloric restriction in humans: impact on physiological, psychological, and behavioral outcomes. Antioxid Redox Signal. 2011 Jan 15;14(2):275-87. doi: 10.1089/ars.2010.3253. Epub 2010 Aug 28. PMID 20518700
- [Background] Fontana L, Partridge L, Longo VD. Extending healthy life span--from yeast to humans. Science. 2010 Apr 16;328(5976):321-6. doi: 10.1126/science.1172539. PMID 20395504
- [Background] Henning SM, Shao P, Qing-Yi L, Yang J, Huang J, Ru-Po L, Thames G, Heber D, Li Z. Health effects of 3-day fruit and vegetable juice fasting. Advanced Nutrition, 7(48A), 2016.
- [Background] Rink SM, Mendola P, Mumford SL, Poudrier JK, Browne RW, Wactawski-Wende J, Perkins NJ, Schisterman EF. Self-report of fruit and vegetable intake that meets the 5 a day recommendation is associated with reduced levels of oxidative stress biomarkers and increased levels of antioxidant defense in premenopausal women. J Acad Nutr Diet. 2013 Jun;113(6):776-85. doi: 10.1016/j.jand.2013.01.019. Epub 2013 Mar 19. PMID 23522825
- [Background] Zheng J, Zhou Y, Li S, Zhang P, Zhou T, Xu DP, Li HB. Effects and Mechanisms of Fruit and Vegetable Juices on Cardiovascular Diseases. Int J Mol Sci. 2017 Mar 4;18(3):555. doi: 10.3390/ijms18030555. PMID 28273863

DOCUMENTS (2):
  • Informed Consent Form (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03647449/ICF_000.pdf
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03647449/Prot_001.pdf